CLINICAL TRIAL: NCT05851352
Title: Predictive Value of Serum Anti-endometrial Antibodies in Implantation Rate for Patient With Endometriosis Undergoing Intracytoplasmic Sperm Injection Cycles
Brief Title: anti_endometrial Antibodies in Endometriosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammed Zain Al_a'bdeen, doctor, South Valley University
Other Study IDs: anti_endometrial antibodies
Record Dates: First submitted 2023-05-01; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Anti-endometrial Antibodies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum anti-endometrial antibodies — - Take blood samples from patients to measure anti-endometrial antibody concentrations in the serum of women with endometriosis using human Endometrium Antibody, EMAb ELISA Kit .This assay employs the qualitative enzyme immunoassay technique

SUMMARY:
The aims of this study is to asses the predictive value of serum anti_endometrial antibodies in prediction of implantation rate in patient with endometriosis who undergoing intracytoplasmic sperm injection cycles.

DETAILED DESCRIPTION:
prospective cohort study of infertile patients ( with endometriosis & adenomyosis) who will undergo ICSI cycles at the assisted reproduction units,Obstetrics and Gynacology departments , South Valley University and Cairo University.

Initial evaluation: this will include:

1. Detailed history and clinical examination.
2. Ovarian reserve testing (serum AMH , basal serum FSH and basal AFC by US)
3. Uterine cavity examination ( by trasvaginal 3-dimentional ultrasound or office hysteroscopy)
4. routine investigations (Complete blood count, blood grouping , liver function tests , kidney function tests , prothrombin time , prothrombin concentration , serum bloog sugar)
5. Evaluation of male factor (husbnad semen analysis)

   * Eligible women will undergo :

     * Transvaginal ultrasound for evaluation of endometriosis ( shape , size , unilateral or bilateral , unilocular or bilocular )
     * Perform laparscopy for confirmation of endometriosis using revised ASM classification for endometriosis
     * Measurement of serum anti_endometrial antibodies :
     * Take blood samples from patients to measure anti-endometrial antibody concentrations in the serum of women with endometriosis using human Endometrium Antibody, EMAb ELISA Kit .

Intracytoplasmic sperm injection (ICSI) gonadotrophin stimulation drugs will be used, individualization of stimulation dose and slight modifications will be done according to ovarian response. Proper protocol will be used. Baseline assessment of AFC by transvaginal scans wasill be performed by experienced gynaecologist using a 7.5 MHz vaginal probe 7-MHz (Samsung, Korea). Ovarian response monitoring to stimulation drug, estimation the doses of gonadotrophins required for follicular growing and maturation, assessment the stimulation time in days till time of ovum pick-up, and the number and quality of oocytes obtained will be recorded in and analysed at the end of the study. When 3-4 follicles acquired >18 mm ,triggering of ovulation will be done using human chorionic gonadotrophins 36 hours prior to pick-up of oocytes. after oocyte retrieval ICSI procedure will be done for all cases. embryos will be transferred to each mother on day 3 or day 5 according to embryos quality and remaining of good quality embryos will be frozen for subsequent transfer. Luteal support started in day of ova pick up till date of pregnancy test (14 days post embryos transfer)

Research outcome measures:

a. Primary (main):

* assess the predictive value of serum antiendometrial antibodies in prediction of implantation rate in patient with endometriosis who undergoing intracytoplasmic sperm injection cycles b. Secondary (subsidiary):
* to find correlation between serum anti-endometrial antibodies and egg quality retrieved

ELIGIBILITY:
Inclusion Criteria:

- Patients will be enrolled in this study if they fulfill the following criteria:

1. infertile patients (with endometriosis & adenomyosis ) who will undergo ICSI cycles
2. Age: 18-35 years.
3. Body mass index (BMI): ≤ 30.
4. primary or secondary infirtility. 5 duration of infertility less than 10 years

6. results of semen examination of patients' husbands will be within the World Health Organization (WHO) reference range.

Exclusion Criteria:

Patients will not be eligible for this study if:

1. gynecological problem e.g. uterine polyp, hydrosalpinx will be excluded 2. Male factor: Abnormal sperm morphology;(globozoospermia and pin- point sperm) will be excluded 3 . congenital structural abnormalities of the reproductive tract, pelvic tuberculosis, ovarian tumour, hyperprolactinaemia, adrenal disease, thyroid disease or other endocrine disease,

-

Ages: 15 Years to 35 Years | Sex: Female
Age Groups: Child, Adult
Study Population: infertile patients ( with endometriosis & adenomyosis) who will undergo ICSI cycles at the assisted reproduction units,Obstetrics and Gynacology departments , South Valley University and Cairo University.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
serum antiendometrial antibodies and implantation rate in patient with endometriosis who undergoing intracytoplasmic sperm injection cycles | baseline
  assess the predictive value of serum antiendometrial antibodies in prediction of implantation rate in patient with endometriosis who undergoing intracytoplasmic sperm injection cycles

SECONDARY OUTCOMES:
serum antiendometrial antibodies in patient with endometriosis who undergoing intracytoplasmic sperm injection cycles and egg quality retrieved | baseline
  find correlation between serum anti-endometrial antibodies and egg quality retrieved

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahman A Elsayed, professor, Study Chair — South Valley University; mostafa M Khodry, lecturer, Study Chair — South Valley University; Radwa M Fahmy, lecturer, Study Chair — Cairo University
Locations (1):
- Mohammed Zain Al_a'bdeen, Qina, Maabar, Egypt

REFERENCES:
- [Background] Giudice LC, Kao LC. Endometriosis. Lancet. 2004 Nov 13-19;364(9447):1789-99. doi: 10.1016/S0140-6736(04)17403-5. PMID 15541453
- [Background] Hummelshoj L, Prentice A, Groothuis P. Update on endometriosis. Womens Health (Lond). 2006 Jan;2(1):53-6. doi: 10.2217/17455057.2.1.53. No abstract available. PMID 19803926
- [Background] Geva E, Amit A, Lerner-Geva L, Lessing JB. Autoimmunity and reproduction. Fertil Steril. 1997 Apr;67(4):599-611. doi: 10.1016/s0015-0282(97)81351-9. PMID 9093180
- [Background] Choudhury SR, Knapp LA. Human reproductive failure I: immunological factors. Hum Reprod Update. 2001 Mar-Apr;7(2):113-34. doi: 10.1093/humupd/7.2.113. PMID 11284658
- [Background] Palacio JR, Iborra A, Ulcova-Gallova Z, Badia R, Martinez P. The presence of antibodies to oxidative modified proteins in serum from polycystic ovary syndrome patients. Clin Exp Immunol. 2006 May;144(2):217-22. doi: 10.1111/j.1365-2249.2006.03061.x. PMID 16634794
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/14885276/